CLINICAL TRIAL: NCT00464958
Title: Long Term Clinical Efficacy and Safety of Novel Sublingual Tizanidine HCl (12 mg) for the Treatment of Spasticity in Patients With Multiple Sclerosis - Open Label Extension Study
Brief Title: One Year Extension Study To Protocol C2/5/TZ:MS-05
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was stopped as the sponsor is no longer funding this project
Sponsor: Teva GTC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol C2/5/TZ:MS-05 EXT
Record Dates: First submitted 2007-04-22; First posted 2007-04-24 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-01

CONDITIONS: Spasticity; Multiple Sclerosis
Keywords: Fatigue; Spasticity; Sublingual Tizanidine; Epworth Sleepiness Scale; Fatigue Severity Scale
MeSH Terms: conditions — Muscle Spasticity; Multiple Sclerosis; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sublingual tizanidine (Experimental): Once nightly dosing of 12 mg sublingual tizanidine tablet
  Interventions: Drug: sublingual tizanidine 12 mg

INTERVENTIONS:
Drug: sublingual tizanidine 12 mg — Single sublingual tizanidine 12 mg tablet, to be administered once nightly, via sublingual administration for 12 months

SUMMARY:
Open label, one year extension study to evaluate the clinical efficacy and safety of 12 mg sublingual tizanidine administered once nightly in MS patients who successfully completed Phase I/II protocol C2/5/TZ:MS-05 at the Tel Aviv Sourasky Medical Center, Department of Neurology, Dr. Arnon Karni, PI.

DETAILED DESCRIPTION:
The previous study, Protocol C2/5/TZ-MS-05, using 12 mg sublingual tizanidine, confirmed that administration of once nightly sublingual tizanidine before sleep results in a statistically and clinically significant reduction in next-day spasticity, as compared to placebo. The clinical effect following 12 mg sublingual tizanidine was larger (4-5 units on the Ashworth scale) and more sustained (up to 18-20 hours post-dose) than was seen for 8 mg tizanidine (earlier study, Protocol C2/5/TZ:MS-03z). This study also reconfirmed that the increased improvement in next-day reduction of spasticity following overnight sublingual tizanidine dosing is not accompanied by a concomitant increase in next-day somnolence.

This study, a 12 month open label extension, will allow those patients who successfully completed Protocol C2/5/TZ-MS-05 and who found tizanidine to be beneficial, to continue treatment under close medical supervision. The study will provide long-term (12 months) clinical efficacy and safety data re: the use of once daily sublingual tizanidine, administered at night, just before bedtime.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of previous protocol, Study C2/5/TZ:MS-05
* Have a definitive diagnosis of Multiple Sclerosis
* Patients may be allowed to take other anti-spasticity medication during the study (other than Baclofen pump)as per their individual daily dosing regimen, with the following qualification: (1) No dose after 18:00 on any study day (2) No dose at all on a clinic evaluation day
* Females must agree to use a medically accepted form of birth control, be surgically sterile, or be two years post-menopausal. Oral contraception in NOT acceptable as it is contraindicated for tizanidine use.
* Patients must meet criteria for stable 24 hour BP values based on the screening ABPM monitorings (with and without tizanidine challenge) as determined by the study's BP consultant

Exclusion Criteria:

* Use of CYP1A2 inhibitors [e.g. ciprofloxacin or fluvoxamine as well as zileuton, other fluroquinolones (norfloxacin), antiarrythmics (amiodarone, mexiletine, propafenone), cimetidine, famotidine, oral contraceptives, acyclovir, and ticlopidine] from baseline and for the duration of the study
* Taking medications from baseline and for the duration of the study that would potentially interfere with the actions of the study medication or outcome variables as determined by the PI
* Previous history of dementia, unstable psychiatric disease or current signs and symptoms of significant medical disorders such as severe, progressive or uncontrolled renal, hepatic hematological, endocrine, pulmonary, cardiac, neurological or cerebral disease
* Significant abnormalities in screening laboratory parameters as described below:
* ALT > 2xULN
* AST > 2xULN
* Creatinine > 2.0 mg/dL
* Bilirubin > 2xULN
* WBC < 2,300/mm3
* Platelets < 80,000/mm3
* History of allergy to tizanidine or any inactive component (including lactose intolerance) of the sublingual tizanidine tablet
* History of substance abuse within past 12 months
* Patients who are non-cooperative or unwilling to sign consent form

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Clinical Efficacy- reduction in next-day spasticity (Ashworth scores) | 12 months
Safety- No increase in next-day somnolence/fatigue, measured via Epworth Sleepiness Scale (ESS) and Fatigue Severity Scale (FSS) questionnaires | 12 months

SECONDARY OUTCOMES:
Additional Safety Measures: Clinical Laboratories (hematology and clinical chemistry, with special emphasis on liver function tests); Blood pressure monitoring (standard vital signs: BP and pulse at every monthly visit, + 24 hour Holter ambulatory Blood | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Karni, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- See also: ClinicalTrials.gov Identifier: NCT00358293 — http://www.clinicaltrials.gov/ct2/results?term=NCT00358293